CLINICAL TRIAL: NCT04031066
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Velmanase Alfa in Patients With Alpha Mannosidosis
Brief Title: Interventional Study to Assess Efficacy and Safety of Velmanase Alfa in Patients With Alpha Mannosidosis
Acronym: SHAMAN
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Big delay on study activation (approval procedures by IRBs, hospitals contract negotiation) and on enrolment deadline due to CoViD-19; Placebo stock expires November 2021 and new batch not be available for at least one year
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-LMZYMAA2-01
Record Dates: First submitted 2019-07-17; First posted 2019-07-24 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Alpha-Mannosidosis
Keywords: Alpha-Mannosidosis; velmanase alfa; alpha-mann; shaman; mannosidosis; alpha-mannosidasis
MeSH Terms: conditions — alpha-Mannosidosis; Mannosidase Deficiency Diseases

STUDY DESIGN:
Intervention Model Description: double-blind, randomized 2:1 to either velmanase alfa:placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized using IRT system
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Velmanase alfa (Experimental)
  Interventions: Drug: Velmanase Alfa
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Velmanase Alfa — infusion i.v. treatment
  Arms: Velmanase alfa
Drug: Placebo — infusion i.v. treatment
  Arms: placebo

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel group study where subjects will receive velmanase alfa or placebo for 24 weeks.

Each subject undergoes to 8 complete visits at the clinic for clinical, laboratory and functional assessments. Study treatment is administered weekly through i.v. infusions

DETAILED DESCRIPTION:
A Screening visit (V1) will take place 7±3 days prior to randomization in order to give the subject enough time to consider their participation in the study, to plan the next visits including the long-stay visits at V2, V5 and V8 (long-stay visits as PK and certain tests are performed over more than one day), and to allow the clinic center to complete the evaluation of the eligibility criteria.

Upon confirmation of eligibility, subjects will be randomized to receive weekly i.v. administration of either velmanase alfa 1 mg/kg or placebo.

Thereafter, subjects will undergo weekly visits for administration of study treatment and safety data collection. Clinical, laboratory and functional assessments will be performed at the 4-weekly assessment visits with each subject undergoing a minimum of 8 assessment visits (V1 to V8).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of alpha-mannosidosis based on alpha mannosidase activity <10% of normal in leukocytes or fibroblasts or through genetic testing;
* Capability to comply with the protocol;
* Evidence of informed consent provided by subject or legally authorized guardian(s) prior to performance of any trial-related activities.

Exclusion Criteria:

* Previous hematopoietic stem cells transplantation (HSCT) with positive outcome;
* Major surgery planned within 3 months prior to study entry or planned during the study that, in the opinion of the Investigator, would preclude participation in the trial;
* Known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical condition that would preclude participation in the study in the Investigator's judgment;
* Pregnant (as evident by a positive urine hCG or serum-hCG test) or lactating women and all women physiologically capable of becoming pregnant (i.e. women of childbearing potential [WOCBP]) UNLESS they are willing to use highly effective birth control methods;
* Participation in other interventional trials testing investigational medicinal products (IMPs) within the last 6 months;
* Total IgE >800 IU/ml;
* Any hypersensitivity to velmanase alfa or its excipients that, in the judgment of the Investigator, places the subject at an increased risk for adverse reactions
* Clinically active infection and recent vaccinations (within the last month before screening).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-11 (Estimated); Primary Completion 2021-10-27 (Estimated); Study Completion 2021-12-29 (Estimated)

PRIMARY OUTCOMES:
Change in concentration of serum oligosaccharides | 24 weeks (end of study)
  To evaluate the efficacy of velmanase alfa compared with placebo after 24 weeks of velmanase alfa treatment as measured by Level of serum oligosaccharides;
Change in serum level of total immunoglobulin (Ig)G level | 24 weeks (end of study)
  Efficacy of velmanase alfa compared with placebo in alpha mannosidosis subjects based on serum levels of total immunoglobulin (Ig)G after 24 weeks of velmanase alfa treatment

SECONDARY OUTCOMES:
Change in Intracellular level of oligosaccharides in peripheral blood leukocytes | 24 weeks (end of study)
  To evaluate the efficacy of velmanase alfa compared with placebo after 24 weeks of velmanase alfa treatment as measured by Intracellular level of oligosaccharides accumulated in peripheral blood leukocytes.
Change in serum IgG Subclasses | 24 weeks (end of study)
  To evaluate the efficacy of velmanase alfa compared with placebo after 24 weeks of velmanase alfa treatment as measured by Subclasses of IgG;
Incidence of Infections | 24 weeks (end of study)
  Change in number of infections requiring antibiotics and/or hospitalization and/or loss of school/working days
Assessment of PK parameter Maximum plasma Concentration [Cmax] | 12 weeks
  To collect additional data on Cmax profile following velmanase alfa treatment
Assessment of PK parameter Maximum plasma Concentration [Cmax] | 24 weeks (end of study)
  To collect additional data on Cmax profile following velmanase alfa treatment
Assessment of PK parameter Area Under the Curve [AUC] | 24 weeks (end of study)
  To collect additional data on AUC profile following velmanase alfa treatment
Assessment of PK parameter Area Under the Curve [AUC] | 12 weeks
  To collect additional data on AUC profile following velmanase alfa treatment
Assessment of PK parameter Elimination half-life [t1/2] | 12 weeks
  To collect additional data on t1/2 profile following velmanase alfa treatment
Assessment of PK parameter Elimination half-life [t1/2] | 24 weeks (end of study)
  To collect additional data on t1/2 profile following velmanase alfa treatment
Assessment of PK parameter trough concentration (Ctrough) | 12 weeks
  To collect additional data on Ctrough profile following velmanase alfa treatment
Assessment of PK parameter trough concentration (Ctrough) | 24 weeks (end of study)
  To collect additional data on Ctrough profile following velmanase alfa treatment

OTHER OUTCOMES:
Adverse Events (AEs) | 24 weeks (end of study)
  Number of AEs will be described for each patient and cumulatively in the safety population
Infusion Related Reactions (IRRs) | 24 weeks (end of study)
  Number of IRRs will be described for each patient and cumulatively in the safety population
Incidence of Adverse Drug Reactions (ADRs) | 24 weeks (end of study)
  Number of ADRs will be described for each patient and cumulatively in the safety population
Anty-Drug Antibody (ADA) level | 24 weeks (end of study)
  Change in ADA will be described for each patient and cumulatively in the safety population
Neutralizing Antibody (NAb) level | 24 weeks (end of study)
  Change in NAb levels will be described for each patient and cumulatively in the safety population
Change on Immunoglobuline Type A (IgA) values | 24 weeks (end of study)
  Change in IgA levels will be described for each patient and cumulatively in the safety population
Change on Immunoglobuline Type M (IgM) values | 24 weeks (end of study)
  Change in IgM levels will be described for each patient and cumulatively in the safety population
Change on B-cell immunophenotype level | 24 weeks (end of study)
  Change in B-cell immunophenotype levels will be described for each patient and cumulatively in the safety population
3MSCT (3-Minute Stair Climb Test) | 24 weeks (end of study)
  Change from baseline in motricity tests (climbing test) will be described for each patient
6MWT (2MWT for children) (6- or 2-Minute Walk Test) | 24 weeks (end of study)
  Change from baseline in motricity tests (walking test) will be described for each patient
FVC, FEV1 and PEF | 24 weeks (end of study)
  Change from baseline in respiratory tests (Spirometry) will be described for each patient
Psychotic events | 24 weeks (end of study)
  Change from baseline in number of psychotic events will be described for each patient
Shoulder mobility | 24 weeks (end of study)
  Change from baseline in shoulder mobility will be described for each patient
ECG PR interval | 24 weeks (end of study)
  Change from baseline in electrocardiogram (ECG) PR interval will be described for each patient
ECG QT interval | 24 weeks (end of study)
  Change from baseline in electrocardiogram (ECG) QT interval will be described for each patient
ECG QRS duration | 24 weeks (end of study)
  Change from baseline in electrocardiogram (ECG) QRS duration will be described for each patient
Heart diseases | 24 weeks (end of study)
  Change from baseline in Echocardiogram will be described for each patient
Hearing testing | 24 weeks (end of study)
  Change from baseline in hearing testing through PTA will be described for each patient
Kaufman-II (Kaurfman Assessment Battery for Children - 2nd Edition) | 24 weeks (end of study)
  Change in score from baseline in cognitive testing Kaufman-II will be described for each patient
Bayley-III (Bayley Scales of Infant and Toddler Development - 3rd Edition) | 24 weeks (end of study)
  Change in score from baseline in cognitive testing Bayley-III will be described for each patient
VABS-3 scores (Vineland Adaptive Behavior Scales - 3rd Edition) | 24 weeks (end of study)
  Change in score from baseline in cognitive testing VABS-3 will be described for each patient
Development Motor scale | 24 weeks (end of study)
  Change from baseline in Peabody Delelopment Motor scale (PMDS-2) scores will be described for each patient
EQ-5D-5L (European Quality of Life Five Dimension Five Level) Questionnaire | 24 weeks (end of study)
  Change in score from baseline for questionnaire EQ-5D-5L will be described for each patient
CHAQ (Childhood Health Assessment Questionnaire) | 24 weeks (end of study)
  Change in score from baseline for CHAQ will be described for each patient
MPS Health Assessment Questionnaire | 24 weeks (end of study)
  Change in score from baseline for questionnaire MPS Health Assessment Questionnaire will be described for each patient
Zarit Burden Interview | 24 weeks (end of study)
  Change in score from baseline for questionnaire Zarit Burden Interview will be described for each patient
CBCL (Child Behavioral Checklist) or ABCL (Adult Behavioral Checklist) according to age | 24 weeks (end of study)
  Change in score from baseline for CBCL or ABCL will be described for each patient
PEDI (Pediatric Evaluation of Disability Inventory) | 24 weeks (end of study)
  Change in score from baseline for PEDI will be described for each patient
PROMIS-SF (Patient-reported Outcomes Measurement Information System Short Forms) | 24 weeks (end of study)
  Change in score from baseline for PROMIS-SF will be described for each patient
Service-use and cost questionnaire to patient and families | 24 weeks (end of study)
  Change in score from baseline will be described for each patient
Physician's Judgement of Overall Response | 24 weeks (end of study)
  Change from baseline based on a Likert scale (0 to 5)
Caregiver's Judgement of Overall Response | 24 weeks (end of study)
  Change from baseline based on a Likert scale (0 to 5)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Harmatz, MD, Principal Investigator — UCSF Benioff Children's Hospital Oakland

IPD SHARING:
Plan to Share IPD: No